CLINICAL TRIAL: NCT05028257
Title: Pursuit of Vaccination in Anaphylactic Reaction to COVID19 Vaccines
Brief Title: Allergy and COVID-19 Vaccines
Acronym: COVALL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 210641; 2021-003155-42 (EudraCT Number)
Record Dates: First submitted 2021-07-31; First posted 2021-08-31 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Anaphylactic Reaction; Vaccine Reaction
Keywords: Anaphylactic reactions; COVID-19 vaccines; PEG2000; tromethamine
MeSH Terms: conditions — Anaphylaxis | interventions — COVID-19 Vaccines; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COVID-19 Vaccinated Patients (Experimental)
  Interventions: Biological: COVID-19 Vaccines

INTERVENTIONS:
Biological: COVID-19 Vaccines — Pursuit of vaccination in case of anaphylactic reaction
  Other Names: Janssen COVID19 vaccine; Astra Zeneca COVID19 vaccine; Comirnaty Pfizer COVID19 vaccine; Moderna COVID19 vaccine

SUMMARY:
Prospective and retrospective multicenter study to estimate the proportion of patients who tolerated continuation of COVID-19 vaccination (absence of anaphylactic manifestations).

secondly, to determine the proportion of definite anaphylactic reactions in cases of suspected anaphylaxis following administration of a COVID-19 vaccine.

Comprehensive allergological investigations involving clinical, skin and biological tests will enable us to determine whether or not vaccine components, and in particular excipients (PEG2000, PS80 and tromethamine), are responsible for anaphylactic reactions to COVID-19 vaccines.

A biological collection will be set up during this clinical study to study the immunological mechanisms, effector cells and signalling pathways involved in these reactions.

DETAILED DESCRIPTION:
Eligible patients will be identified via the pharmacovigilance centers and allergology hotlines set up in each center, according to the organization specific to each hospital site. .

The patient identified in this way will be contacted by the secretariat of each allergology center to schedule an allergology consultation at least 3 to 5 weeks after the reaction (the usual delay before exploring an anaphylactic reaction to avoid the risk of false negatives). Then, in the framework of a collegial meeting ,the patient's file will be reviewed in order to specify the history of the allergic disease and the modalities of subsequent COVID-19 vaccination.

A follow-up telephonique call at 6months will be made systematically for patients who have continued vaccination to ensure that there are no significant adverse events related to the COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Anaphylactic reaction to a COVID-19 vaccine administered by Pfizer-BioNtech or Janssen or Vaxzevria or Moderna, at least 3 weeks old at the time of the allergology consultation.

An anaphylactic reaction is defined as the occurrence of any of the following systemic manifestations within a few hours of administration of a COVID-19 vaccine:

* skin rash with urticaria and/or angiodema,
* and/or associated with respiratory signs (dyspnea, bronchospasm, desaturation), and/or digestive disorders (intense abdominal pain, diarrhea, vomiting, nausea), and/or neurological disorders (loss of consciousness, feeling of malaise), and/or hypotension, tachycardia.
* Affiliation to a Social Security system
* Signature of the informed consent
* Stop taking antihistamines at least 3 days before skin allergy tests are performed

Exclusion Criteria:

* Other non-anaphylactic systemic reactions after administration of COVID-19 mRNA vaccine (serum sickness, vasculitis, Guillain-Barré syndrome)
* Pregnancy and lactation
* Disorders of hemostasis or severe bleeding considered a contraindication to intramuscular injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Describe the continuation of vaccination and its tolerance in case of negative allergological investigation. | from Week 9 to Month 9
  Proportion of patient without anaphylactic reaction during second vaccination

SECONDARY OUTCOMES:
Determine the involvement of excipients in anaphylactic reactions | from Week 9 to Month 9
  Proportion of patient with positive skin tests for excipients (PEG2000, PS80) or COVID-19 vaccines
To determine with certainty the diagnosis of anaphylaxis in the face of a suspected anaphylactic reaction during the administration of a COVID-19 vaccine. | from Week 9 to Month 9
  Proportion of patient with positive allergological explorations (anamnesis, skin tests or biological test for excipients or vaccines)

CONTACTS AND LOCATIONS:
Overall Officials: Angèle SORIA, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Tenon Hospital APHP dermatology and allergology department, Paris, France

IPD SHARING:
Plan to Share IPD: No